CLINICAL TRIAL: NCT06790199
Title: A Mixed-methods Evaluation of the Implementation of a Teacher Classroom Program to Support Preschool Children With Autism or Developmental Problems: A Feasibility Randomized Controlled Pilot Trial
Brief Title: Implementation of a Teacher Classroom Program to Support Preschool Children With Autism or Developmental Problems
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-179-24
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder; Teacher Training; Teacher Skills in Addressing Child Mental Health Problem; Developmental Disorders
Keywords: Autism; Teacher training; Developmental disorders; Randomized controlled trial; Early intervention; Mental health
MeSH Terms: conditions — Autism Spectrum Disorder; Developmental Disabilities; Autistic Disorder; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Incredible Years-Helping Preschool Children with Autism program) (Experimental): Teachers in the intervention group will receive the Incredible Years-Helping Preschool Children with Autism program (IY-HPCA).
  They will participate in a 6-session group-based face-to-face intervention. Sessions will last 3 hours, will be delivered weekly at Hospital Sant Joan de Déu, and will be led by two trained co-leaders. The following main topics will be covered: (1) language development, (2) social interactions, and (3) emotion literacy and self-regulation.
  Two groups will be conducted, and each of them will include around 10 teachers.
  Interventions: Behavioral: Incredible Years® "Helping Preschool Children with Autism" program (IY-HPCA)
- Control group (No Intervention): The control group will not receive the intervention. Teachers who are assigned to the control group will continue their usual teaching practice.
  No restrictions will be placed on schools regarding access to other training and support services during the course of the study, but this information will be monitored as a potential confounder.
  Teachers who are assigned to the intervention group will be asked not to share the intervention contents with other teachers who are in the control group before the end of the study.

INTERVENTIONS:
Behavioral: Incredible Years® "Helping Preschool Children with Autism" program (IY-HPCA) — The IY-HPCA® program is a face-to-face 6-session group-based intervention for preschool teachers of children aged 2-5 with ASD or language and communication difficulties. Sessions last 3 hours, are delivered weekly, and are led by two trained co-leaders who have experience working with children on the autism spectrum. The program covers three main topics: (1) language development, (2) social interactions, and (3) emotion literacy and self-regulation. Teachers learn about coaching language, imitation, sensory routines, social communication, use of pretend and puppet play, and self-regulation skills. Visual supports such as picture schedules, choice cards, command and feelings cards are used, and practices are tailored to children's communication and play level stages. The intervention is structured and includes role-playing techniques and video visualization.
  Arms: Intervention group (Incredible Years-Helping Preschool Children with Autism program)

SUMMARY:
The Incredible Years® "Helping Preschool Children with Autism" (IY-HPCA) program is designed for teachers of children aged 2 to 5 years who have students with autism in their classrooms. The program provides tools to support children with autism.

The primary aim of this pilot study is to examine the feasibility of implementing the IY-HPCA intervention among teachers of preschool children (typically aged 2 to 5 years) working in mainstream schools. Specifically, the study aims to assess teachers' engagement, acceptability, and satisfaction with the program. Secondarily, it aims to gather preliminary evidence on the program's effectiveness in improving teachers' use of strategies, teacher self-efficacy, and in reducing burnout.

An exploratory randomized controlled pilot trial will be conducted. Approximately 40 teachers will be recruited, and they will be randomly assigned to either an intervention or control group.

The intervention consists of six weekly sessions lasting 3 hours each, delivered by clinical psychologists and child psychiatrists specialized in developmental disorders at Hospital Sant Joan de Déu, in Barcelona. Two intervention face-to-face groups will be conducted at Hospital Sant Joan de Déu.

Feasibility outcomes include program attendance, acceptability, and satisfaction (assessed using the Incredible Years Teacher Workshop Evaluations and the Teacher Satisfaction Questionnaire), as well as fidelity to the intervention delivery (measured with the Leader Checklist). After the intervention, individual interviews with teachers and group leaders will qualitatively assess satisfaction and experiences with the program.

Secondary (effectiveness) outcomes include teachers' use of strategies (Teacher Strategies Questionnaire for Children with Autism), self-efficacy (Teacher Sense of Efficacy Scale), and burnout (Maslach Burnout Inventory-Educators Survey).

This study will provide pioneering insights into the implementation of this program within the public mental health and education systems in Spain. This will allow the potential implementation of a wider randomized controlled trial in the future at a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Teachers working at mainstream schools near the catchment area of Hospital Sant Joan de Déu Barcelona.
* Teachers working at mainstream schools with specific programs for children with special needs.
* Teachers of pre-school children.
* Teachers willing to participate in the study and signing the inform consent.

Exclusion Criteria:

- Teachers working at special education centers instead of mainstream schools.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of teachers engaging with and finishing the program | Attendance sheet completed weekly throughout the intervention (6 weeks total)
  Teachers' attendance at the sessions will be regeristered weekly with a sheet of attendance, with the aim to determine levels of compliance and engagement with the intervention. An attendance of at least 4/6 sessions is expected, with a minimum of 50% of teachers finishing the program.
Compliance and satisfaction throughout the study (Incredible Years Teacher Weekly Evaluations) | Questionnaire administered to the intervention group weekly throughout the intervention (6 weeks total)
  Teachers' compliance and satisfaction with the intervention will be assessed weekly after each session with the questionnaire "Incredible Years Teacher Weekly Evaluations", which is part of the IY-HPCA® program materials.
  This weekly assessment asks teachers to rate their satisfaction with different aspects of the program.
Teachers' acceptability and satisfaction with the program (evaluated with the Final Participant Satisfaction Questionnaire) | Administered to the intervention group at intervention completion (approximately 6 weeks after baseline)
  Teachers' acceptability and satisfaction with the program will be assessed with the Final Participant Satisfaction Questionnaire-Helping Preschool Children with Autism Program (included within the IY-HPCA® program). Data will be collected after the last session of the intervention.
Teachers' overall experiences with the program (evaluated with individual interviews) | Interviews to the participants of the intervention group at intervention completion (approximately 6 weeks after baseline)
  Individual interviews will be conducted after the last session of the intervention to explore from a qualitative perspective: (1) teachers' acceptability, satisfaction and overall experience and perceptions of the intervention, and (2) teachers' perceived changes in their skills after the intervention.
  Outcome measurements 3 and 4 will be combined to determine teachers' experiences, acceptability and satisfaction with the program.
Group leaders' fidelity with the program (evaluated with the Leader Checklist) | Leader Checklist completed weekly throughout the intervention (6 weeks total)
  Fidelity with the program will be assessed weekly after each session with the "Leader Checklist", which is part of the IY-HPCA® program materials. Group leaders (clinicians) will complete the Leader Checklist.
Clinicians' experiences with the intervention delivered (evaluated with individual interviews) | Interviews to clinicians at intervention completion (approximately 6 weeks after baseline)
  Individual interviews will be conducted after the last session with clinicians who delivered the intervention.

SECONDARY OUTCOMES:
Changes from baseline to post-intervention in Teacher Strategies Questionnaire for Children with Autism (TSQ-A) | Administered to the intervention and control group at baseline (prior to programme initiation) and after the intervention (approximately 6 weeks after baseline)
  The Teacher Strategies Questionnaire for Children with Autism (TSQ-A) is a 52-item teacher-report questionnaire part of the IY program materials that consists of six sections. The first section asks teachers to rate their confidence in promoting social, emotional, language and academic development of children with ASD. Sections 2-4 ask teachers to rate the frequency with which they use teaching techniques to support children's language, social and emotional development. In the last section, teachers rate the frequency of their planning and support strategies according to a five-point scale.
Changes from baseline to post-intervention in Teacher Sense of Efficacy Scale-Long Version | Administered to the intervention and control group at baseline (prior to programme initiation) and after the intervention (approximately 6 weeks after baseline)
  The Teacher Sense of Efficacy Scale-Long Version (Tschannen-Moran & Hoy, 2001; Spanish version: Salas-Rodríguez et al., 2021) is a 24-item questionnaire that measures teachers' evaluations of how likely they are to be successful in teaching. Three different subscales are differentiated: efficacy for classroom management, efficacy to promote student engagement, and efficacy in using instructional strategies.
Changes from baseline to post-intervention in Maslach Burnout Inventory-Educators Survey | Administered to the intervention and control group at baseline (prior to programme initiation) and after the intervention (approximately 6 weeks after baseline)
  The Maslach Burnout Inventory-Educators Survey (Maslach et al., 1986) is a version of the original Maslach Burnout Inventory for use with educators, including teachers, and has three scales that examine the three core aspects of burnout: emotional exhaustion (feelings of being emotionally overextended and exhausted by one's work), depersonalization (unfeeling and impersonal response toward recipients of one's instruction) and personal accomplishment (feelings of competence and successful achievement in one's work with students).

CONTACTS AND LOCATIONS:
Locations (1):
- Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hayes R, Titheradge D, Allen K, Allwood M, Byford S, Edwards V, Hansford L, Longdon B, Norman S, Norwich B, Russell AE, Price A, Ukoumunne OC, Ford T. The Incredible Years(R) Teacher Classroom Management programme and its impact on teachers' professional self-efficacy, work-related stress, and general well-being: Results from the STARS randomized controlled trial. Br J Educ Psychol. 2020 May;90(2):330-348. doi: 10.1111/bjep.12284. Epub 2019 Apr 13. PMID 30980389
- [Background] Serrano M, Elias M, Llorens M, Bolasell M, Vall-Roque H, Villalta L. Early treatment for children with mental health problems and genetic conditions through a parenting intervention (The GAP): study protocol for a pragmatic randomized controlled trial. Trials. 2024 Jul 20;25(1):496. doi: 10.1186/s13063-024-08278-4. PMID 39033111
- See also: Information on The Incredible Years teacher programs — https://www.incredibleyears.com/training/prepare#teacher